CLINICAL TRIAL: NCT02398097
Title: Safety and Immunogenicity of Influenza Vaccine Among HIV-infected Young Subjects: Conventional Vaccine Versus Intradermal Vaccine
Brief Title: Conventional Vaccine and Intradermal Vaccine Among HIV-infected Young Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hee Jin Cheong, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLUHIV
Record Dates: First submitted 2015-03-01; First posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Human Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Agripal (Active Comparator): 28 trivalent subunit inactivated intramuscular vaccine (Agripal) recipients: one vaccine injection administered on Day 0
  Interventions: Biological: Agripal
- IDflu9μg (Active Comparator): 30 reduced-content intradermal split vaccine (IDflu9μg) recipients: one vaccine injection administered on Day 0
  Interventions: Biological: IDflu9μg
- IDflu15μg (Active Comparator): 28 standard-content intradermal split vaccine (IDflu15μg) recipients: one vaccine injection administered on Day 0
  Interventions: Biological: IDflu15μg

INTERVENTIONS:
Biological: Agripal — 2011/2012 influenza season standard dose trivalent subunit inactivated intramuscular vaccine, single dose
  Arms: Agripal
Biological: IDflu9μg — 2011/2012 influenza season reduced-content intradermal split vaccine, single dose
  Arms: IDflu9μg
Biological: IDflu15μg — 2011/2012 influenza season standard-content intradermal split vaccine, single dose
  Arms: IDflu15μg

SUMMARY:
Several studies have shown poor immune response to conventional influenza vaccines in HIV-infected individuals. This study was conducted expecting the more potent immunogenicity of intradermal vaccine compared with conventional intramuscular vaccine in HIV-infected adults.

DETAILED DESCRIPTION:
During the 2011/2012 pre-influenza season, three vaccines were used in HIV-infected adults (18 to 60 years): inactivated intramuscular vaccine (Agripal), reduced-content intradermal vaccine (IDflu9μg) and standard-content intradermal vaccine (IDflu15μg). Serum hemagglutination-inhibiting (HI) antibodies and INF-γ ELISpot assay were measured at the time of vaccination and 1 month after vaccination. Adverse events were recorded for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individuals who were not immunized with 2011/2012 influenza vaccine

Exclusion Criteria:

* known allergy to egg
* presentation of any febrile illness ≥37.5°C on the day of vaccination
* any history of hypersensitivity reaction to previous influenza vaccination
* any other vaccinations within the past one month
* use of immunosuppressive agent
* recipient of blood product or immunoglobulins during the previous three months
* any other conditions that might interfere with the study results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with a post-vaccination titer ≥1:40 in subjects with a pre-vaccination titer of <1:10 or a ≥4-fold titer increase in subjects with a pre-vaccination titer of ≥1:10 | Outcome measure was assessed at two points (baseline and 4 weeks after vaccination)

SECONDARY OUTCOMES:
Percentage of subjects with a post-vaccination titer ≥1:40 | Outcome measure was assessed 4 weeks after vaccination
GMT ratio of the post-vaccination titer to pre-vaccination titer | Outcome measure was assessed at two points (baseline and 4 weeks after vaccination)

OTHER OUTCOMES:
Frequency and duration of local and systemic adverse events | Adverse events were recorded for 7 days.
  The diary was made based on the Food and Drug Association (FDA) Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jin Cheong, MD, PhD, Principal Investigator — Korea University Guro Hospital

REFERENCES:
- [Derived] Seo YB, Lee J, Song JY, Choi HJ, Cheong HJ, Kim WJ. Safety and immunogenicity of influenza vaccine among HIV-infected adults: Conventional vaccine vs. intradermal vaccine. Hum Vaccin Immunother. 2016;12(2):478-84. doi: 10.1080/21645515.2015.1076599. PMID 26431466